CLINICAL TRIAL: NCT04393870
Title: Effect of Focusing on Maryam's Flower During the First Phase of the Labor
Brief Title: Focusing on Maryam's Flower at Labor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Balikesir University (Other)
Responsible Party: Principal Investigator, Hülya TÜRKMEN, Lecturer (PhD), Balikesir University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: BalıkesirH
Record Dates: First submitted 2020-05-11; First posted 2020-05-19 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Labor Pain; Satisfaction
Keywords: comfort at labor; labor pain; Maryam's flower; focused attention; birth satisfaction
MeSH Terms: conditions — Labor Pain; Personal Satisfaction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Maryam's Flower Group (Experimental): Maryam's flower was placed in a bowl of water and left in the room of the pregnant women who were at 1 cm cervical dilatation and in the first phase of the labor. It was explained to the pregnant women that the leaves of the plant would open up in the water, and they were asked to imagine that the birth canal would simultaneously open up. In effect, they were told to focus on the opening of these leaves during the course of the labor
  Interventions: Other: Foccusing on Maryam's Flower
- Control Group (No Intervention): All the pregnant women, those in the control group, were provided with standard midwifery care.

INTERVENTIONS:
Other: Foccusing on Maryam's Flower — Effect of Focusing on Maryam's Flower During the First Phase of the labor
  Arms: Maryam's Flower Group

SUMMARY:
Objective: To determine the effect that focusing attention on the plant, Maryam's Flower, has on pregnant women's perception of pain, level of comfort and labor satisfaction during the first phase of labor.

Method: This randomized controlled experimental study was conducted with an intervention group (n=61) and control group (n=63) involving primipara pregnant women who were at 1 cm cervical dilatation. The pregnant women in the intervention group were asked to focus their attention on Maryam's flower opening its leaf buds and imagine the labor's progress during the course of their labor. The control group only received standard midwifery care. Each group was administered the VAS at specific times (at 4-5 cm, 6-7 cm, and 8-9 cm cervical dilatation) to determine their level of labor pain. The Childbirth Comfort Questionnaire (CCQ) was also administered when the women were at 4-5 cm and 8-9 cm cervical dilatation to determine their level of birth comfort. The duration of labor was monitored using a partograph form. Finally, the Birth Satisfaction Scale was applied to determine the women's satisfaction with the labor in the 2nd hour of the postpartum period.

DETAILED DESCRIPTION:
Design and Settings This randomized controlled experimental study was conducted in the delivery room of the Atatürk City Hospital in Balıkesir, Turkey between the dates of May 2019 and January 2020.

Participants The sample size was determined using G * Power 3 power calculations, taking into consideration previous studies on the effect of positive mental imagination during labor. Impact predictions were obtained from the findings derived from Yavari et al., which specified the pain intensity during 6-7 cm cervical dilatation to be 6.73 ± 1.34 in the positive mental imagination group, and 7.63 ± 1.64 in the control group (18). This study expected to detect differences similar to those reported by Yavari et al. The sample size was determined to be 61 for each group. Maryam's flower group included 61 pregnant women, while the control group included 63 pregnant women. In the Maryam's flower group, 6 pregnant women and in the control group, 2 pregnant women underwent cesarean sections, therefore, the study was completed with 55 pregnant women from the Maryam's flower group and 61 pregnant women from the control group (The pregnant women underwent cesarean sections after 6-7 cm cervical dilatation). The power analysis indicated that the sample size of the study had a power of 94% with α = 0.05. The decrease observed in labor pain for the Maryam's flower group at 6-7 cm cervical dilatation had an effect size of 0.59 when compared to the control group.

Study inclusion criteria included pregnant women who expected vaginal delivery and a single healthy fetus, who were primipara and in the first phase of the labor, and who were at 1 cm cervical dilatation. Pregnant women who were multipara, had a risky pregnancy, a child with complications, multiple pregnancies, or a premature delivery and those who delivered after 1 cm cervical dilatation were excluded from the study.

Single-blind block randomization was performed with closed opaque envelopes, where 61 of the 124 envelopes include pieces of paper on which were written "intervention" and 63 on which were written "control". The randomization sequence was determined by a statistician through a computerized research randomizer. The intervention group focused on Maryam's flower throughout the delivery, while the control group was provided standard midwifery care.

Data Collection The participating pregnant women who were in the first phase of labor and at 1 cm cervical dilatation were administered an introductory information form. In the intervention group, Maryam's flower was placed in a bowl of water once the women were at 1 cm cervical dilatation, and the pregnant women were asked to focus on the plant. Each group, that is, the intervention group and the control group, were administered the Visual Analog Scale (VAS-1) when they were at 4-5 cm cervical dilatation and the Childbirth Comfort Questionnaire, to detect their levels of birth comfort, and the VAS-2 when they were at 6-7 cm cervical dilatation. Once the women reached 8-10 cm cervical dilation, they were asked to respond to the VAS-3 and Childbirth Comfort Questionnaire. The Birth Satisfaction Scale was used to determine the level of postnatal satisfaction.

Measures The study data were collected through the Pregnant Information Form, the VAS, the Partograph form, the Childbirth Comfort Questionnaire, and the Birth Satisfaction Scale.

The Pregnant Information Form (PIF): This form included questions on the sociodemographic, gynecological, and obstetric characteristics of the pregnant women.

Visual Analog Scale (VAS): This scale was used to determine the level of labor pain. The scale features a 10-cm long vertical line, with 0 at the bottom end and 10 at the top end. The VAS was administered when the women were at 4-5 cm, 6-7 cm, and 8-10 cm cervical dilatation, and the women completed the scale themselves Partograph Form: This form was used to determine the duration of the first phase of the labor process (active phase and transition phase).

Childbirth Comfort Questionnaire (CCQ): This questionnaire was developed by Kerri Durnell Schuling and Carolyn Sampselle in 2003 (7). The Turkish reliability and validity study of the questionnaire was conducted by Potur et al. (2015) (11), who reported that the CCQ included physical, environmental, and psychospiritual subscales and relief and transcendence levels. The questionnaire features 9 items, each of which are evaluated based on a 5-point Likert-type scale, where 1 represented strongly disagree and 5 represented strongly agree. The minimum and maximum scores possible on the scale are 9 and 45, respectively, with higher scores representing higher levels of comfort and lower scores representing lower levels. Potur et al. found Cronbach's alpha reliability coefficient to be 0.75. The CCQ was administered twice in this study, once at 4-5 cm cervical dilatation and once at 8-9 cm cervical dilatation.

The Birth Satisfaction Scale (BSS): The Turkish reliability and validity study of this scale developed by Hollins Martin and Fleming was conducted by Çoşar et al. (2015). The scale is a Likert-type scale comprised of 30 questions. The minimum and maximum scores possible on the scale are 30 and 150, respectively. Higher scores indicate higher birth satisfaction. An analysis conducted to determine the internal consistency of the BSS found the Cronbach's alpha value to be 0.62. The BSS was administered at the 2nd hour of the postnatal period.

Intervention Maryam's flower was placed in a bowl of water and left in the room of the pregnant women who were at 1 cm cervical dilatation and in the first phase of the labor. It was explained to the pregnant women that the leaves of the plant would open up in the water, and they were asked to imagine that the birth canal would simultaneously open up. In effect, they were told to focus on the opening of these leaves during the course of the labor (Pictures 1 and 2). All the pregnant women, those in the control group and in intervention group, were provided with standard midwifery care. As part of the standard midwifery care given to the pregnant women, follow-up of cervical dilatation and effacement, contraction, fetal heart rate, and vital signs were monitored. The pregnant women were given information on breathing and pushing techniques. Moreover, induction was performed on all the pregnant women. in labor.

ELIGIBILITY:
Inclusion Criteria:

* expected vaginal delivery
* single healthy fetus
* primipara
* in the first phase of the labor
* 1 cm cervical dilatation

Exclusion Criteria:

* multipara
* risky pregnancy
* child with complications
* multiple pregnancies
* premature delivery
* after 1 cm cervical dilatation

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnant women
Enrollment: 124 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
severity of labor pain by VAS | immediately after the intervention
  Visual Analog Scale The scale features a 10-cm long vertical line, with 0 at the bottom end and 10 at the top end
duration of active phase and transition phase of labor (4-10cm cervical dilatation) | during the procedure
  duration of active phase and transition phase of labor (4-10cm cervical dilatation)
comfort level at labor | immediately after the intervention
  Childbirth Comfort Questionnaire (CCQ) 5-point Likert-type- minimum 9 and maximum 45 points are obtained from the scale. higher scores mean a better comfort

SECONDARY OUTCOMES:
birth satisfaction level. | 2nd hour of the postnatal period.
  The Birth Satisfaction Scale, Likert-type scale- minimum 30 and maximum 150 points are obtained from the scale. higher scores mean a better birth satisfaction

CONTACTS AND LOCATIONS:
Locations (1):
- Hülya TÜRKMEN, Balıkesir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Turkmen H, Cetinkaya S, Kilic H, Apay E, Karamuftuoglu D, Yoruk S, Ozkirim E. Effect of Focusing on Maryam's Flower During the First Stage of the Labor on the Labor Pain, Labor Duration, and Levels of Comfort and Satisfaction. Clin Nurs Res. 2021 Jul;30(6):780-789. doi: 10.1177/1054773820984911. Epub 2020 Dec 29. PMID 33371726